CLINICAL TRIAL: NCT02332044
Title: A Randomized, Open-label, Single Dose, Three-treatment, Three-period, Six-sequence Crossover Study to Investigate the Pharmacokinetic Drug Interaction Between Erdosteine and Bepotastine Besilate After Oral Administration in Healthy Volunteers
Brief Title: Drug Interaction Study Between Erdosteine and Bepotastine Besilate in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW_DWJ1340001
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Erdosteine 300mg (Experimental)
  Interventions: Drug: Erdos
- Bepotastine besilate 10mg (Experimental)
  Interventions: Drug: Talion
- Erdosteine 300mg + Bepotastine besilate 10mg (Experimental)
  Interventions: Drug: Erdos, Talion

INTERVENTIONS:
Drug: Erdos — capsule, 300mg
  Arms: Erdosteine 300mg
Drug: Talion — tablet, 10mg
  Arms: Bepotastine besilate 10mg
Drug: Erdos, Talion — capsule 300mg and tablet 10mg
  Arms: Erdosteine 300mg + Bepotastine besilate 10mg

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction between Erdosteine and Bepotastine besilate in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 45 years
* A body mass index in the range 18.5 - 25 kg/m2
* Willingness to participate during the entire study period
* Written informed consent after being fully informed about the study procedures

Exclusion Criteria:

* Any past medical history of hepatic, renal, gastrointestinal, respiratory, endocrine, psychiatric, neurologic, haemato-oncologic or cardiovascular disease
* History of clinically significant drug hypersensitivity
* Use of medication within 7 days before the first dose
* Heavy drinker/smoker
* Whole blood donation during 60 days before the study
* Judged not eligible for study participation by investigator

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cmax | Multiple blood sample will be collected for 24 hours after last dosing in each of the treatment
AUClast | Multiple blood sample will be collected for 24 hours after last dosing in each of the treatment